CLINICAL TRIAL: NCT07178054
Title: Total Energy Expenditure in Healthy Chinese Populations: A Nationwide Study Using the Doubly Labelled Water Method
Status: Recruiting | Type: Observational
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Xueying Zhang, Associate researcher, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Other Study IDs: SIAT-IRB-250815-H1005
Record Dates: First submitted 2025-08-25; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples will be collected from children and adults over a 14-day period following the administration of doubly labelled water (DLW). The analysis of oxygen-18 and deuterium in these urine samples will be used to calculate the total energy expenditure of the children and the adults.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Between 1990 and 2022, the global prevalence of obesity more than doubled, representing a critical public health concern. China has mirrored this trend, with rapidly increasing rates of overweight and obesity across all age groups. According to the 'Report on Chinese Residents' Nutrition and Chronic Diseases (2020)', 50.7% of Chinese adults are now classified as overweight or obese. Among children and adolescents aged 6 to 17 years, data from the 'Atlas of Nutrition and Health Status of Chinese Children' indicates that the prevalence of overweight and obesity has reached 26.5%.

Obesity is associated with a broad spectrum of adverse health outcomes across the life course. In children, excess adiposity negatively affects skeletal maturation, neurocognitive development, and psychosocial well-being, while also increasing the likelihood of obesity and metabolic dysfunction in adulthood. In adults, obesity is a major risk factor for a range of non-communicable diseases (NCDs), including type 2 diabetes mellitus, hypertension, cardiovascular disease, non-alcoholic fatty liver disease, osteoarthritis, certain cancers, and all-cause premature mortality. Beyond its health implications, obesity imposes substantial economic and social burdens, including increased healthcare expenditure and reduced workforce productivity.

The etiology of the obesity epidemic is multifactorial and remains under active investigation. Hypotheses center around a chronic imbalance between energy intake and expenditure, driven by behavioral, environmental, and physiological factors. Notably, decreased physical activity associated with sedentary lifestyles and increased consumption of energy-dense, nutrient-poor foods have been implicated as key contributors. However, the relative contributions of reduced energy expenditure versus increased energy intake remain insufficiently quantified at the population level. Accurate assessment of total energy expenditure (TEE) is therefore essential to elucidate the energy dynamics underlying the obesity epidemic.

Current approaches for estimating population-level energy and food requirements are often based on indirect methods with limited precision. The doubly labelled water (DLW) technique, which quantifies TEE through measurement of isotope elimination rates (^2H and ^18O), remains the gold standard for assessing free-living energy expenditure. However, its application has been predominantly confined to high-income countries with well-established research infrastructure. In contrast, the use of DLW in low- and middle-income countries-including China-remains minimal, resulting in critical data gaps that hinder the development of context-specific dietary recommendations and energy requirement models.

To address these limitations, this study will apply the DLW method to measure TEE in healthy children and adults in China. In parallel, the study will assess key modulators of energy metabolism, including anthropometric and physiological parameters, gut microbiota composition, habitual physical activity, and ambient temperature exposure. The resulting dataset will provide high-resolution, population-specific evidence to inform national dietary reference intakes and support the formulation of evidence-based public health strategies aimed at obesity prevention and metabolic health promotion.

DETAILED DESCRIPTION:
The investigators will recruit healthy children aged 7 to 18 and healthy adults aged 30 to 60 from within the country to participate in a study to explore their energy requirements and factors.

The following measurements will be conducted in both children and adults:

1. Study Details Anthropometric Measurements

   1. Height: Height will be measured using a Seca 217 stadiometer. Participants will stand barefoot with feet approximately 60° apart. Heels, sacrum, and shoulder blades will be placed against the stadiometer's vertical rod. The head will be aligned so that the upper margin of the ear canal is level with the lower margin of the eye socket. The horizontal plate will be lowered gently to rest on the crown of the head. Two measurements will be taken and averaged; values will be recorded to the nearest 0.1 cm.
   2. Body Weight: After an overnight fast, body weight will be measured in the morning using a calibrated TANITA MC-780 scale. Participants will wear light clothing and no shoes.
   3. Waist Circumference: Waist circumference will be measured at the midpoint between the iliac crest and the lower edge of the 12th rib. Participants will stand with feet 25-30 cm apart and body weight evenly distributed. A flexible tape will be wrapped snugly (without compression), and two measurements will be averaged to the nearest 0.1 cm.
   4. Hip Circumference: Hip circumference will be measured with the participant standing straight, legs together, arms relaxed. The tape will be placed horizontally at the level of the pubic symphysis and the most prominent part of the buttocks. Two measurements will be taken and averaged.
   5. Thigh Circumference: Thigh circumference will be measured with the participant standing straight, legs together, arms relaxed. The tape measure should be wrapped horizontally around the thickest part of the thigh (usually about 10 centimeters below the hip crease), closely adhering to the skin but not pressing on the soft tissue. The average of two measurements will be taken, accurate to 0.1 cm.
   6. Neck Circumference: Neck circumference will be measured with the participant keeping their head straight and drooping their shoulders naturally. The tape measure should be placed horizontally at the lower edge of the thyroid cartilage (Adam's apple) in front of the neck, passing through the lower part of the bilateral occipital protuberances on both sides. The measurement should be taken twice and the average value will be obtained, accurate to 0.1 cm.
   7. Blood Pressure: Blood pressure will be measured with the participant relaxing shoulders, straightening backs, sitting upright and placing arms flat on the table at the same level as the heart. Participants will rest quietly for more than 5-10 minutes before measuring blood pressure. The blood pressure cuff will tie at a distance of one finger above the elbow, with the center point level with the heart. Record the blood pressure at the end.
   8. Heart Rate: Heart rate will be measured with the participant relaxing shoulders, straightening backs, sitting upright and placing arms flat on the table at the same level as the heart. Participants will rest quietly for more than 5-10 minutes before measuring blood pressure. The blood pressure cuff will tie at a distance of one finger above the elbow, with the center point level with the heart. Record the heart rate at the end.
   9. Abdominal Fat: Abdominal fat will be measured with the participant lying on their back and exposing abdomen as instructed by the doctor. Trained personnel will use the DW-360 to measure participants' abdominal fat.
   10. Bone Mineral Density: Bone mineral density will be measured with the participant lying flat on their back and remaining still as instructed by the technician. Professional personnel will use the Dual Energy X-ray (DXA) scanner to measure participants' bone mineral density.
2. Blood biochemistry test and gut microbiota detection

   1. Blood Index: Blood index will be measured by taking blood samples from participants after a 10-hour fast, including red blood cell (RBC), white blood cells (WBC), hemoglobin (HB), etc.
   2. Lipid Profile: Lipid profile will be measured by taking blood samples from participants after a 10-hour fast, including total cholesterol, triglycerides, high-density lipoprotein cholesterol (HDL-C) and low-density lipoprotein cholesterol (LDL-C).
   3. Liver Function: Liver function will be measured by taking blood samples from participants after a 10-hour fast, including alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TB), direct bilirubin (DB) and indirect bilirubin (IB), etc.
   4. Renal Function: Renal function will be measured by taking blood samples from participants after a 10-hour fast, including blood urea nitrogen (BUN), serum uric acid (SUA) and serum creatinine (SCr).
   5. Vitamin D levels: Vitamin D levels will be measured by taking blood samples from non-fasting participants.
   6. Gut Microbiota: Gut microbiota is obtained by collecting fecal samples from participants.
3. Questionnaires

   1. Comprehensive questionnaire for adults: Will be conducted through a set of questionnaires covering demographic information, past health conditions, dietary structure, and sleep quality.
   2. Pubertal development for children under guardianship: Will be assessed via Tanner staging for secondary sexual characteristics.
   3. Dietary intake for participants: Will be assessed using three 24-hour dietary recall questionnaires administered on non-consecutive days.
4. Body composition and energy expenditure

   1. Body Composition:

      Bioelectrical impedance analysis (TANITA MC-780) and DXA (Hologic, Horizon Wi)will be used to measure segmental weight (arms, legs, trunk), total body fat percentage (fat%), fat mass (FM), fat-free mass (FFM), total body water (TBW) and muscle mass.
   2. Basal Metabolic Rate(BMR) :

      Basal metabolic rate will be measured using indirect calorimetry via a Cosmed Quark system with a ventilated hood. After a 10-hour overnight fast and no strenuous activity in the preceding day, participants will lie supine under the hood for 30 minutes. Oxygen consumption and carbon dioxide production will be monitored, and the final 10 minutes will be used to calculate BMR (Weir, 1949). Equipment will be validated monthly via alcohol burn tests and turbine flow calibration.
   3. Total Energy Expenditure:

      Total energy expenditure (TEE) will be measured using the doubly labelled water (DLW) method. Urine samples will be collected and stored at -20°C, then shipped on dry ice to Dr. John Speakman's laboratory at the University of Aberdeen or to the Shenzhen Institute of Advanced Technology. Isotope ratios will be analyzed using a near-infrared isotope gas analyzer. Mean CO2 production will be calculated using equations developed by Speakman et al. (2021), and TEE will be derived using the Weir equation (1949).
   4. Environmental Temperature Exposure:

      Environmental temperature exposure will be monitored using iButton sensors (DS1921G). These will be placed in the participant's living environment (eg, on a backpack, clothing, indoor wall, or building exterior) using waterproof medical-grade adhesive. This will allow measurement of ambient temperature during the study period.
   5. Physical Activity:

Physical activity will be monitored using ActiGraph GT3X accelerometers worn at the waist for 14 consecutive days, except during water activities (e.g., bathing or swimming). Data will be considered valid if the monitor is worn for at least 12 hours on four days, including at least two weekdays and two weekend days. The first day of wear and any day with insufficient data will be excluded from analysis.

The following additional measurements will be performed in children:

1. Mid-Upper Arm Circumference: Mid-upper arm circumference will be measured with the participant standing straight, legs together, arms relaxed. The midpoint between the acromion (shoulder) and olecranon (elbow) will be marked. A measuring tape will be wrapped around this midpoint with light contact. Two measurements will be taken and averaged.
2. Grip Strength: Grip strength will be measured by the dynamometer(CAMRY, EH101), Read the displayed number on the dynamometer as the grip strength value. Take the maximum value of the two measurements, accurate to 0.1 kg.
3. Skin Carotenoid: Skin carotenoid will be measured with the participant covering the non-index finger on the veggie meter. The non-index finger will clean with alcohol to ensure they were free of oil and fat before measuring. Then, the content of carotenoids in the participant's skin will be accurately evaluated.

This study will provide accurate data on the energy consumption of healthy people living in China. These data will serve as a basis for estimating the country's food and energy requirements, support public health nutrition strategies, and help fill the key data gaps in the domestic DLW database.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants

Exclusion Criteria:

* Exclusion Criteria:

  1. Malnutrient as defined by the Chinese national standards WS/T456-2014 and WS/T 586-2018

     1. Nutritional deficiencies
     2. Overweight
     3. Obesity
  2. Acute illness within the past 7 days

     1. Fever
     2. Diarrhea
     3. Vomiting
  3. Chronic diseases

     1. Cardiovascular diseases
     2. Diabetes mellitus or any form of metabolic disorders

        * Type 1 or Type 2 diabetes
        * Metabolic syndrome
        * Hyperlipidemia
        * Dyslipidemia
     3. Renal diseases

        * Chronic kidney disease
        * Nephrotic syndrome
  4. Musculoskeletal injuries
  5. Disabilities

Ages: 7 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The research participants will consist of healthy adults aged 30 to 60 and healthy children aged 7 to 18 years who exhibit normal growth and development. All participants are neither overweight nor obese, nor will they have any nutritional deficiencies. They will be capable of cooperating to complete all necessary measurements. None of these participants has been diagnosed with chronic diseases, musculoskeletal injuries or disabilities. Moreover, all participants will be free from acute clinical diseases at least seven days prior to the study.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Height | About 3 minutes.
  Height in meters will be measured by Leicester stadiometer (Seca 217, Germany) and reported to two decimal places.
Weight | About 5 minutes.
  Weight in kilograms will be measured by TANITA.
BMI | About 10 minutes (calculated)
  BMI values in kg/m2 will be calculated from weight measured by TANITA and height measured by Leicester stadiometer (Seca 217, Germany).
Fat mass | About 3 minutes.
  Fat mass in kilograms will be measured by TANITA.
Fat percentage | About 3 minutes.
  Fat percentage will be measured by TANITA.
Fat-free mass | About 3 minutes.
  Fat-free mass in kilograms will be measured by TANITA.
Muscle mass | About 3 minutes.
  Muscle mass in kilograms will be measured by TANITA.
Total body water | About 3 minutes.
  Total body water in kilograms will be measured by TANITA.
Waist circumference | About 5 minutes.
  Waist circumference(measured in centimeters) will be obtained using a flexible tape measure following standardized protocols.
Hip circumference | About 5 minutes.
  Hip circumference(measured in centimeters) will be obtained using a flexible tape measure following standardized protocols.
Thigh circumference | About 5 minutes.
  Thigh circumference(measured in centimeters) will be obtained using a flexible tape measure following standardized protocols.
Neck circumference | About 5 minutes.
  Neck circumference(measured in centimeters) will be obtained using a flexible tape measure following standardized protocols.
Blood pressure | About 10 minutes.
  Blood pressure will be measured using a standardized blood pressure monitor, with recordings of both systolic and diastolic values.
Heart rate | About 10 minutes.
  Heart rate will be measured in using a standardized blood pressure monitor.
Abdominal fat | About 20 minutes.
  Abdominal fat will be measured in using a portable ultrasound device (DW-360).
Bone mineral density | About 20 minutes.
  Bone mineral density will be measured using the Dual-energy X-ray Absorptiometry (DXA) device.
Mid-upper arm circumference | About 5 minutes.
  Mid-upper arm circumference (measured in centimeters) will be obtained using a flexible tape measure following standardized protocols.
Grip strength | About 5 minutes.
  Grip strength will be obtained using a dynamometer(CAMRY, EH101).
Skin carotenoid concentration | About 5 minutes.
  Skin carotenoid concentration will be measured in using the Veggie Meter，and the results will be expressed as Standard Point Score (SPS), typically ranging from 0 to 800 SPS. Higher SPS values indicate higher skin carotenoid concentration.
Red Blood Cell Count | About 10 minutes.
  Red blood cell count will be measured in fasting blood samples.
White Blood Cell Count | About 10 minutes.
  White blood cell count will be measured in fasting blood samples.
Hemoglobin | About 10 minutes.
  Hemoglobin concentration will be measured in fasting blood samples, reported in grams per liter (g/L).
Total Cholesterol | About 10 minutes.
  Total cholesterol concentration will be measured in fasting blood samples, reported in millimoles per liter (mmol/L).
Triglycerides | About 10 minutes.
  Triglycerides concentration will be measured in fasting blood samples, reported in millimoles per liter (mmol/L).
High-Density Lipoprotein Cholesterol | About 10 minutes.
  High-density lipoprotein cholesterol (HDL-C) concentration will be measured in fasting blood samples, reported in millimoles per liter (mmol/L).
Low-Density Lipoprotein Cholesterol | About 10 minutes.
  Low-density lipoprotein cholesterol (LDL-C) concentration will be measured in fasting blood samples, reported in millimoles per liter (mmol/L).
Alanine Aminotransferase | About 10 minutes.
  Alanine aminotransferase (ALT) activity will be measured in fasting blood samples, reported in units per liter (U/L).
Aspartate Aminotransferase | About 10 minutes.
  Aspartate aminotransferase (AST) activity will be measured in fasting blood samples, reported in units per liter (U/L).
Total Bilirubin | About 10 minutes.
  Total bilirubin concentration will be measured in fasting blood samples, reported in micromoles per liter (μmol/L).
Direct Bilirubin | About 10 minutes.
  Direct bilirubin concentration will be measured in fasting blood samples, reported in micromoles per liter (μmol/L).
Indirect Bilirubin | About 10 minutes.
  Indirect bilirubin concentration will be measured in fasting blood samples, reported in micromoles per liter (μmol/L).
Blood Urea Nitrogen | About 10 minutes.
  Blood urea nitrogen (BUN) concentration will be measured in fasting blood samples, reported in millimoles per liter (mmol/L).
Serum Uric Acid | About 10 minutes.
  Serum uric acid concentration will be measured in fasting blood samples, reported in micromoles per liter (μmol/L).
Serum Creatinine | About 10 minutes.
  Serum creatinine concentration will be measured in fasting blood samples, reported in micromoles per liter (μmol/L).
Vitamin D levels | About 10 minutes.
  Vitamin D levels will be obtained by collecting blood samples.
Gut microbiota | About 10 minutes.
  Gut microbiota will be obtained by collecting fecal samples.
Secondary sexual characteristics | About 5 minutes.
  The Tanner stages are used to assess the development of secondary sexual characteristics and are divided into five stages. For boys, the evaluation includes pubic hair development and genital development (including testicular and penile growth). For girls, the evaluation includes pubic hair development and breast development (thelarche).
Basal metabolic rate | About 30 minutes.
  The basal metabolic rate in kcal or MJ will be measured by respiratory indirect calorimetry (Cosmed).
Total energy expenditure | About 14 days.
  Total energy expenditure in kcal or MJ will be measured using the DLW method. TEE will then be calculated using mean CO2 production using the Weir equation.
Environmental temperature | About 14 days.
  The iButton (DS1921G) monitors will be provided for the assessment of both indoor and outdoor temperature of their living environment, measured in degrees Celsius (°C).
Physical activity energy expenditure | About 14 days.
  Physical activity energy expenditure will be recorded using a GT3X accelerometer worn at the waist for a consecutive period of 14 days, with results expressed in kilocalories (kcal) or megajoules (MJ) per day.
Total moderate-to-vigorous physical activity (MVPA) | About 14 days.
  Total MVPA will be recorded using a GT3X accelerometer worn at the waist for a consecutive period of 14 days, with results expressed in minutes per day (min/day).
Vector magnitude counts | About 14 days.
  Vector magnitude counts will be recorded using a GT3X accelerometer worn at the waist for a consecutive period of 14 days, with results expressed as counts per minute (cpm). Higher cpm values indicate greater overall physical activity intensity, reflecting the average level of movement during the monitoring period.

CONTACTS AND LOCATIONS:
Overall Officials: Xueying Zhang, PhD, Principal Investigator — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (7):
- China (7):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Shenzhen Institutes of Advanced Technology,Chinese Academy of Sciences, Shenzhen, Guangdong
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Qingdao Center Hospital of Rehabilitation University, Qingdao, Shandong
  - Tacheng Prefecture People's Hospital, Tacheng, Xinjiang

REFERENCES:
- [Background] Speakman JR, Yamada Y, Sagayama H, Berman ESF, Ainslie PN, Andersen LF, Anderson LJ, Arab L, Baddou I, Bedu-Addo K, Blaak EE, Blanc S, Bonomi AG, Bouten CVC, Bovet P, Buchowski MS, Butte NF, Camps SGJA, Close GL, Cooper JA, Creasy SA, Das SK, Cooper R, Dugas LR, Ebbeling CB, Ekelund U, Entringer S, Forrester T, Fudge BW, Goris AH, Gurven M, Hambly C, El Hamdouchi A, Hoos MB, Hu S, Joonas N, Joosen AM, Katzmarzyk P, Kempen KP, Kimura M, Kraus WE, Kushner RF, Lambert EV, Leonard WR, Lessan N, Ludwig DS, Martin CK, Medin AC, Meijer EP, Morehen JC, Morton JP, Neuhouser ML, Nicklas TA, Ojiambo RM, Pietilainen KH, Pitsiladis YP, Plange-Rhule J, Plasqui G, Prentice RL, Rabinovich RA, Racette SB, Raichlen DA, Ravussin E, Reynolds RM, Roberts SB, Schuit AJ, Sjodin AM, Stice E, Urlacher SS, Valenti G, Van Etten LM, Van Mil EA, Wells JCK, Wilson G, Wood BM, Yanovski J, Yoshida T, Zhang X, Murphy-Alford AJ, Loechl CU, Melanson EL, Luke AH, Pontzer H, Rood J, Schoeller DA, Westerterp KR, Wong WW; IAEA DLW database group. A standard calculation methodology for human doubly labeled water studies. Cell Rep Med. 2021 Feb 16;2(2):100203. doi: 10.1016/j.xcrm.2021.100203. eCollection 2021 Feb 16. PMID 33665639
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301